CLINICAL TRIAL: NCT04266041
Title: High-density EEG in Neurological Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Yinchen Song, Clinical Neurophysiologist, Neuro Diagnostics, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: D18111 30813
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Epilepsy; Tumor; Healthy
Keywords: Electroencephalogram (EEG); Epilepsy; Lesion; Brain; Language; Movement; Sensation; Mapping; Dense-array EEG; High-density EEG; HD-EEG; stroke; Electrical Impedance Tomography
MeSH Terms: conditions — Epilepsy; Neoplasms; Language; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (5):
- High-density EEG localization in epilepsy (Experimental): High-density EEG will be used for brain localization in epilepsy patients
  Interventions: Diagnostic Test: High-density electroencephalogram (HD-EEG)
- High-density EEG localization in healthy controls (Active Comparator): High-density EEG will be used for brain localization in healthy controls
  Interventions: Diagnostic Test: High-density electroencephalogram (HD-EEG)
- High-density EEG localization in tumor patients (Experimental): High-density EEG will be used for brain localization in tumor patients
  Interventions: Diagnostic Test: High-density electroencephalogram (HD-EEG)
- High-density EEG localization in peripheral nerve patients (Experimental): High-density EEG will be used for brain localization in patients with peripheral nerve dysfunction
  Interventions: Diagnostic Test: High-density electroencephalogram (HD-EEG)
- High-density EEG localization in stroke patients (Experimental): High-density EEG will be used for brain localization in patients who have recently experienced a stroke
  Interventions: Diagnostic Test: High-density electroencephalogram (HD-EEG)

INTERVENTIONS:
Diagnostic Test: High-density electroencephalogram (HD-EEG) — This study will focus on obtaining a special type of high-density scalp electroencephalography (HD-EEG) recordings in patients with neurological disorders (i.e., epilepsy, brain tumor, stroke, etc.) and appropriately matched controls. HD-EEG is a scalp EEG which uses up to 256 channels compared to the standard 21 channels used for routine clinical applications. The reason for using more channels to record is for more precise localization of epileptogenic foci and/or more precise mapping of brain functions. This type of EEG requires the use of patient's own MRI scan to precisely localize activity. Therefore, all patients and controls getting an HD-EEG will require a structural MRI scan.

SUMMARY:
The purpose of the study is to use a new method of high-density electroencephalogram (HD-EEG) recording to map brain areas important for movement, sensation, language, emotion, and cognition.

DETAILED DESCRIPTION:
This study will measure brain waves using high-density EEG. Participants will be asked wear a cap with electrodes attached to it. During the recording, participants may be asked to rest, sleep, or complete a task. The tasks involve viewing pictures, answering questions, speaking, or moving an arm or leg. Recordings generally last between 60-120 minutes.*

ELIGIBILITY:
Inclusion Criteria:

* Able to perform the tasks
* Able to give own consent

Exclusion Criteria:

* Any neurologic or psychiatric diagnosis such as stroke, tumor, or psychosis judged to interfere with high-density EEG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-density EEG Localization in Epilepsy | High-density EEG Localization in Healthy Controls | High-density EEG Localization in Tumor Patients | High-density EEG Localization in Peripheral Nerve Patients | High-density EEG Localization in Stroke Patients
Started | 95 | 12 | 1 | 4 | 7
Completed | 95 | 12 | 1 | 4 | 7
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-density EEG Localization in Epilepsy | High-density EEG Localization in Healthy Controls | High-density EEG Localization in Tumor Patients | High-density EEG Localization in Peripheral Nerve Patients | High-density EEG Localization in Stroke Patients | Total
Number analyzed (Participants) | 95 | 12 | 1 | 4 | 7 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: We did not collect age information for the healthy control subjects for the purposes of protecting subjects' personal information.
  years
    number analyzed (Participants) | 95 | 0 | 1 | 4 | 7 | 107
    (all) | 37.55 (13.19) |  | 72 (0) | 42.75 (10.44) | 74.38 (10.42) | 40.59 (16.22)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 patients did the study twice with different subject IDs.
  Participants
    Female | 38 | 3 | 0 | 2 | 1 | 44
    Male | 57 | 9 | 1 | 2 | 6 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 patients did the study twice with different subject IDs.
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 95 | 5 | 1 | 4 | 7 | 112
    Unknown or Not Reported | 0 | 7 | 0 | 0 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 patients did the study twice with different subject IDs.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 1 | 0 | 0 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 1 | 0 | 0 | 0 | 0 | 1
    White | 92 | 4 | 1 | 4 | 7 | 108
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 8 | 0 | 0 | 0 | 9
Region of Enrollment [Number; unit: participants] — Population: 3 patients did the study twice with different subject IDs.
  participants
    United States | 95 | 12 | 1 | 4 | 6 | 119

OUTCOME MEASURES:

1. Primary Outcome: Localizing Brain Regions That Generate Interictal Spikes
Description: The frequency of detecting interictal spikes in HD-EEG The distance between the source location determined by electrical source imaging and the spike locations determined by SEEG studies
Time Frame: From 30-60 min HD-EEG recording, pre-operatively
Population: 95 adult patients were enrolled in this study. Five subjects have already got neurostimulator (RNS or DBS) implanted before the study, of whom the HD-EEG data were excluded for further analysis. Two other subjects' recordings were excluded due to excessive electrical noise or faulty bulk connector. Therefore, 87 subjects with decent resting-state HD-EEG recordings were processed for spike detection. Interictal spikes were detected in the HD-EEG recordings of nearly 60% of subjects (n = 52).
Measure: Count of Participants; unit: Participants
Arm/Group | High-density EEG Localization in Epilepsy
Number analyzed (Participants) | 87
Participants | 52

2. Secondary Outcome: Localize Brain Functions in Patients and Healthy Controls
Description: Localize brain functions using high-density EEG recordings
Time Frame: At baseline for approximately 60 - 90 minutes
Population: healthy control only had sensory and language tasks. Tumor patient only had motor and sensory tasks, also underwent resting-state recording to localize lesion.
  Peripheral nerve patients only had motor and sensory tasks. Stroke patients only had electrical impedance study to localize the lesion.
Measure: Count of Participants; unit: Participants
Arm/Group | High-density EEG Localization in Healthy Controls | High-density EEG Localization in Tumor Patients | High-density EEG Localization in Peripheral Nerve Patients | High-density EEG Localization in Stroke Patients
Number analyzed (Participants) | 12 | 1 | 4 | 7
Participants
  High-gamma for language: number analyzed (Participants) | 12 | 0 | 0 | 0
  High-gamma for language | 12 |  |  |
  Alpha for motor: number analyzed (Participants) | 0 | 1 | 4 | 0
  Alpha for motor |  | 1 | 0 |
  Somatosensory evoked potential: number analyzed (Participants) | 12 | 1 | 4 | 0
  Somatosensory evoked potential | 1 | 1 | 0 |
  Lesion: number analyzed (Participants) | 0 | 1 | 0 | 7
  Lesion |  | 1 |  | 4

3. Secondary Outcome: Localize Brain Areas Involved in Language
Description: Localize brain areas involved in language using high-density EEG recordings
Time Frame: At baseline for approximately 60 - 90 minutes
Population: all normal subjects
Measure: Count of Participants; unit: Participants
Arm/Group | High-density EEG Localization in Healthy Controls
Number analyzed (Participants) | 12
Participants
  Feasible to complete the language task | 12
  high-gamma activity localized to suspected language area | 12

4. Secondary Outcome: Localize Brain Areas Involved in Movement
Description: Localize brain areas involved in movement using high-density EEG recordings
Time Frame: At baseline for approximately 60 - 90 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | High-density EEG Localization in Tumor Patients | High-density EEG Localization in Peripheral Nerve Patients
Number analyzed (Participants) | 1 | 4
Participants
  Tolerated motor task | 1 | 4
  Alpha band activity localized to motor area | 1 | 0

5. Secondary Outcome: Localize Brain Areas Involved in Sensation
Description: Localize brain areas involved in sensation using high-density EEG recordings
Time Frame: At baseline for approximately 60 - 90 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | High-density EEG Localization in Healthy Controls | High-density EEG Localization in Tumor Patients | High-density EEG Localization in Peripheral Nerve Patients
Number analyzed (Participants) | 12 | 1 | 4
Participants
  Tolerated Sensory task | 12 | 1 | 4
  Somatosensory evoked potential captured | 1 | 1 | 0

6. Secondary Outcome: Localize Brain Areas Associated With Lesions
Description: Localize brain areas associated with lesions using high-density EEG recordings
Time Frame: At baseline for approximately 60 - 90 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | High-density EEG Localization in Tumor Patients | High-density EEG Localization in Stroke Patients
Number analyzed (Participants) | 1 | 7
Participants
  Tolerated resting-state recording | 1 | 7
  Abnormality localized | 1 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the consent through the end of participation for each subject (typically one day).
Description: Adverse event collection for each participant was done from the time of consent through the end of study participation.
Arm/Group | High-density EEG Localization in Epilepsy | High-density EEG Localization in Healthy Controls | High-density EEG Localization in Tumor Patients | High-density EEG Localization in Peripheral Nerve Patients | High-density EEG Localization in Stroke Patients
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/12 | 0/1 | 0/4 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/12 | 0/1 | 0/4 | 2/7
Other Adverse Events (participants affected / at risk) | 0/95 | 0/12 | 0/1 | 0/4 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-density EEG Localization in Epilepsy (N=95) | High-density EEG Localization in Healthy Controls (N=12) | High-density EEG Localization in Tumor Patients (N=1) | High-density EEG Localization in Peripheral Nerve Patients (N=4) | High-density EEG Localization in Stroke Patients (N=7)
Death (Vascular disorders) | 0 | 0 | 0 | 0 | 1 — Stroke arm subject was consented and completed one HD-EEG study session. Six days later, the subject was admitted to Palliative Care and died two weeks later of ischemic stroke. The event was assessed to be not related to the study.
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 — Stroke subject was consented and completed one HD-EEG Study session. Four days later, subject made an unsuccessful suicide attempt. Event assessed to be unlikely related to the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-density EEG Localization in Epilepsy (N=95) | High-density EEG Localization in Healthy Controls (N=12) | High-density EEG Localization in Tumor Patients (N=1) | High-density EEG Localization in Peripheral Nerve Patients (N=4) | High-density EEG Localization in Stroke Patients (N=7)
Tingling of left scalp (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) — Stroke subject was consented to the study. During study testing, the subject reported tingling on the left side of their scalp, so the testing was stopped. The tingling was assessed to be probably related to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (6):
  • Study Protocol and Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT04266041/Prot_SAP_000.pdf
  • Informed Consent Form: HD-EEG Informed Consent - Epilepsy (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT04266041/ICF_001.pdf
  • Informed Consent Form: HD-EEG Informed Consent - Healthy Subject (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT04266041/ICF_002.pdf
  • Informed Consent Form: HD-EEG Informed Consent - Peripheral Nerve (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT04266041/ICF_003.pdf
  • Informed Consent Form: HD-EEG Informed Consent - Stroke (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT04266041/ICF_004.pdf
  • Informed Consent Form: HD-EEG Informed Consent - Tumor (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT04266041/ICF_005.pdf